CLINICAL TRIAL: NCT05363189
Title: Optimizing Postoperative Recovery After Breast Reconstruction With Autologous Tissue (BestDIEP)
Acronym: BestDIEP
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-01423-01
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: breast reconstruction; plastic surgery; microsurgery; free flap
MeSH Terms: conditions — Breast Neoplasms | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No venons augmentation: Retrospective group of patients who have not received venous augmentation during their operation.
  Interventions: Procedure: No venous augmentation
- Venous augmentation: Retrospective group of patients who have received venous augmentation during their operation.
  Interventions: Procedure: Venous augmentation
- ERAS protocol: Retrospective group operated according to the traditional ERAS (enhanced recovery after surgery) protocol
  Interventions: Procedure: Traditional ERAS (enhanced recovery after surgery) protocol
- Sahlgrenska recovery protocol: Prospective group operated according to the Sahlgrenska recovery protocol.
  Interventions: Procedure: Sahlgrenska recovery protocol

INTERVENTIONS:
Procedure: Venous augmentation — Increasing the venous drainage of a deep inferior epigastric artery perforator (DIEP) flap by anastomosing the superficial inferior epigastric vein to the cephalic vein
  Other Names: Double venous system drainage; Cephalic vein turndown
  Groups: Venous augmentation
Procedure: Traditional ERAS (enhanced recovery after surgery) protocol — Pre-, peri-, and post-operative care as described in the ERAS protocol
  Groups: ERAS protocol
Procedure: Sahlgrenska recovery protocol — Pre-, peri-, and post-operative care as described in the Sahlgrenska recovery protocol
  Groups: Sahlgrenska recovery protocol
Procedure: No venous augmentation — Traditional deep inferior epigastric artery perforator flap (DIEP)
  Groups: No venons augmentation

SUMMARY:
Women who have their breast reconstructed with autologous tissue seem to be more satisfied with their breast. However, autologous breast reconstruction entails a bigger operation, and the usage of more health care resources, than some other methods, such as implant-based techniques. The main objectives of the present study are to investigate if pre- peri- and postoperative protocols can be safely modified, so the operation demands less resources, while maintaining a low complication rate and a high patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Operated or will be operated with a DIEP flap in the department
* >18 years of age

Exclusion Criteria:

* Inability to leave informed consent
* Inability to understand and speak Swedish (for the questionnaire)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biological women undergoing breast reconstruction with a deep inferior epigastric artery perforator flap in Sahlgrenska university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-operations | 7 days
  Any re-operations performed for any cause during the first 7 days after the operation
Length of stay (LOS) in hospital | 7 days
  Number of days the patient stays in the hospital after the operation

SECONDARY OUTCOMES:
Patient reported satisfaction and quality of life | 12 months
  Measured with BREAST-Q reconstruction. The patient scores different items om a scale and a sum score of 0-100 is calculated for each domain. A higher score indicates a higher satisfaction/quality of life.
Surgical corrections | 5 years
  Number of cosmetic corrections. All types of corrections performed in general or local anesthetics will be included.
Costs | 5 years
  Health economical analysis of direct and indirect cost related to the different protocols

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No